CLINICAL TRIAL: NCT02288234
Title: Telavancin Observational Use Registry (TOUR)
Acronym: TOUR
Status: Completed | Type: Observational
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 0120
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Hospital Acquired Bacterial Pneumonia; Complicated Skin and Skin Structure Infections; Ventilator Associated Bacterial Pneumonia; Gram Positive Infection
Keywords: Registry
MeSH Terms: interventions — telavancin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vibativ: This is an observational study for patients who were already prescribed Vibativ.
  Interventions: Drug: Vibativ

INTERVENTIONS:
Drug: Vibativ — This is an observational study for patients who were already prescribed Vibativ.
  Other Names: telavancin

SUMMARY:
The telavancin observational use registry (TOUR) will collect data to support study of the efficacy, safety, and pattern of use of telavancin in hospital-based inpatients and in outpatients being treated in infusion centers who are receiving clinician directed telavancin therapy.

DETAILED DESCRIPTION:
This is a retrospective medical chart review, multicenter, observational study to examine telavancin efficacy and safety in a real-word setting and to characterize the pattern of use of telavancin in hospital-based inpatients and in outpatient infusion centers. All treatment decisions and clinical assessment will be made at the discretion of the treating physician per usual care and are not mandated by study design or protocol.

ELIGIBILITY:
Inclusion Criteria:

-received at least 1 dose of telavancin since January 1, 2015

Exclusion Criteria:

* Participation in an interventional research study or clinical trial involving telavancin after January 01, 2015

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will aim to enroll approximately 1,000 patients from 50-60 hospital sites or outpatient infusion centers.
Sampling Method: Non-Probability Sample
Enrollment: 1063 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Time to clinical response | 6 months
  defined as the number of days between initiation of telavancin therapy and date of cure, where cure is defined as the resolution of the signs and symptoms of infection and/or no need for additional antibiotic therapy, or clearance of the infection with a negative culture result [Mohr 2009]

SECONDARY OUTCOMES:
Frequency and Proportion of Patients experiencing Renal Adverse Events (AEs) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (1):
- Newland Medical Associates, Southfield, Michigan, United States

REFERENCES:
- [Derived] Sims CR, Bressler AM, Graham DR, Lacy MK, Lombardi DA, Castaneda-Ruiz B. Real-World Clinical Use and Outcomes of Telavancin for the Treatment of Bone and Joint Infections: Results from the Telavancin Observational Use Registry (TOUR). Drugs Real World Outcomes. 2021 Dec;8(4):509-518. doi: 10.1007/s40801-021-00255-6. Epub 2021 May 26. PMID 34041706
- [Derived] Reilly J, Jacobs MA, Friedman B, Cleveland KO, Lombardi DA, Castaneda-Ruiz B. Clinical Experience with Telavancin for the Treatment of Patients with Bacteremia and Endocarditis: Real-World Results from the Telavancin Observational Use Registry (TOUR). Drugs Real World Outcomes. 2020 Sep;7(3):179-189. doi: 10.1007/s40801-020-00191-x. PMID 32372280